CLINICAL TRIAL: NCT04205903
Title: A Phase Ib Study of the Safety and Pharmacology of Nilotinib to Prevent Paclitaxel-Induced Peripheral Neuropathy in Patients With Breast Cancer
Brief Title: Nilotinib in Preventing Paclitaxel-Induced Peripheral Neuropathy in Patients With Stage I-III Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicole Williams, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSU-18317; NCI-2019-03146 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA238946 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-12-20 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — nilotinib; Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15. Patients also receive nilotinib hydrochloride monohydrate PO on days 7, 8, 14, and 15 of cycle 1 and days -1, 1, 7, 8, 14, and 15 of cycle 2. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nilotinib; Drug: Nilotinib Hydrochloride Monohydrate; Drug: Paclitaxel; Other: Questionnaire Administration
- Dose level 2 (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15. Patients also receive nilotinib hydrochloride monohydrate PO on days 7, 8, 14, and 15 of cycle 1 and days -1, 1, 7, 8, 14, and 15 of cycle 2. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nilotinib; Drug: Nilotinib Hydrochloride Monohydrate; Drug: Paclitaxel; Other: Questionnaire Administration
- Dose level 3 (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15. Patients also receive nilotinib hydrochloride monohydrate PO on days 7, 8, 14, and 15 of cycle 1 and days -1, 1, 7, 8, 14, and 15 of cycle 2. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nilotinib; Drug: Nilotinib Hydrochloride Monohydrate; Drug: Paclitaxel; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Nilotinib — Given PO
  Other Names: AMN 107 Base Form
Drug: Nilotinib Hydrochloride Monohydrate — Given PO on cycle 1 Days 7, 14, 15 once a day 24 hours prior to the paclitaxel infusion and again 30 minutes prior to the paclitaxel infusion on days 8, 15.
  Other Names: AMN107; Nilotinib Monohydrochloride Monohydrate; Tasigna
Drug: Paclitaxel — Given IV weekly on days 1, 8, 15, of every 21 days, at a starting dose of 80mg/m2
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase Ib trial studies the side effects and best dose of nilotinib in preventing paclitaxel-induced peripheral neuropathy in stage I-III breast cancer patients who are receiving paclitaxel therapy. Chemotherapy is the usual or standard treatment for breast cancer. It kills cancer cells and lowers the chance that the cancer will come back. Sometimes, this treatment can cause numbness and tingling, especially in the hands and feet. This is called chemotherapy-induced peripheral neuropathy. This study aims to test the safety and effectiveness, both good and bad, of taking nilotinib in preventing chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of nilotinib hydrochloride monohydrate (nilotinib) in combination with paclitaxel.

II. To determine the toxicity profile (based on Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 5.0) of nilotinib in combination with paclitaxel.

SECONDARY OBJECTIVES:

I. To determine the effect of paclitaxel on pharmacokinetics (PK) of nilotinib in the study population.

II. To determine the effect of nilotinib on PK of paclitaxel in the study population.

OUTLINE: This is a phase Ib, dose-escalation study of nilotinib hydrochloride monohydrate.

PHASE Ib: Paclitaxel will be given weekly on days 1, 8, 15, of every 21 days, at a starting dose of 80mg/m2. Nilotinib will be given orally on cycle 1 Days 7, 14 once a day 24 hours prior to the paclitaxel infusion and again 30 minutes prior to the paclitaxel infusion on days 8, 15. During the cycle 1, PK will be obtained at baseline, during, and up to 24 hours after paclitaxel or nilotinib administration on the days 1, 7, 8. Patients will continue paclitaxel without nilotinib after cycle 1 as part of standard of care at the discretion of the treating investigator

ELIGIBILITY:
Inclusion Criteria:

* Men or Women with a known diagnosis of breast cancer stages I-III.
* Be eligible for weekly or dose dense single agent paclitaxel therapy based on physician assessment.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2

  * Patients with ECOG scores of 3 or greater typically do not receive chemotherapeutic intervention.
* Leukocytes >= 2,000/uL.
* Absolute neutrophil count >= 1,500/uL.
* Platelets >= 100,000/uL.
* Total bilirubin =< upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal.
* Creatinine within normal institutional limits OR >= 50 mL/min for patients with creatinine levels above institutional normal.
* Corrected QT interval (QTc) < 450 milliseconds.
* If a female subject is with child bearing potential, she must have a negative pregnancy test at screening.
* Female subjects of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 3 months after completion of study treatment administration. Adequate contraception includes methods such as oral contraceptives, double barrier method (condom plus spermicide or diaphragm), or abstaining from sexual intercourse.
* Be willing and able to understand and sign the written informed consent document.
* Demonstrate adequate electrolyte values as defined below. Hypokalemia and/or hypomagnesemia must be corrected prior to initiating nilotinib:

  * Calcium 8.6-10.5mg/dL
  * Magnesium 1.6-2.6mg/dL

Exclusion Criteria:

* Known distant metastatic disease.
* Is HER2+ and is receiving paclitaxel in conjunction with trastuzumab +/- pertuzumab.
* Has experienced > grade 1 neuropathy during previous therapies for early stage breast cancer.
* Has experienced prior treatment-related toxicities that have not recovered to grade 1 or less (except for alopecia).
* Has a history of grade 3-4 immediate hypersensitivity reaction to paclitaxel.
* Has a history of clinically significant allergic reactions attributed to compounds of similar chemical or biologic composition to nilotinib or paclitaxel.
* Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Is currently pregnant or breast feeding as there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nilotinib and paclitaxel.
* Has any other medical or psychiatric condition that in the opinion of the investigator would make the study therapy unsafe for the patient.
* Has gastrointestinal (GI) disorders or impairment of GI function that is likely to significantly alter the absorption of nilotinib
* Has a marked baseline abnormal heart rhythm such as prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc of > 450msec)
* Has a history of additional risk factors for TdP (e.g., heart failure, hypokalemia, hypomagnesemia, family history of Long QT Syndrome)
* Uses potent CYP3A4 inhibitors (grapefruit juice, cyclosporine, ketoconazole, ritonavir) and if treatment cannot be either safely discontinued or switched to a different medication prior to starting nilotinib.
* Has a known diagnosis of human immunodeficiency virus (HIV) and is currently taking combination antiretroviral therapy known or suspected to affect paclitaxel pharmacokinetics (PK).
* Is concurrently using potent OATP1B1 inhibitors, including antibiotics (rifampicin, rifamycin SV, systemic fusidic acid, clarithromycin, erythromycin, roxithromycin, telithromycin), antiretrovirals (indinavir, saquinavir, ritonavir), cyclosporine, and gemfibrozil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Williams, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stage TB, Hu S, Sparreboom A, Kroetz DL. Role for Drug Transporters in Chemotherapy-Induced Peripheral Neuropathy. Clin Transl Sci. 2021 Mar;14(2):460-467. doi: 10.1111/cts.12915. Epub 2020 Nov 9. PMID 33142018
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven participants enrolled in the study. One participant withdrew prior to be randomized to a dose level,, leaving ten participants who were randomized to the three dose levels.
Groups:
- Dose Level 1 (100mg Nilotinib); Dose Level 2 (200mg Nilotinib); Dose Level 3 (300mg Nilotinib): Patients receive paclitaxel IV on days 1, 8, and 15. Patients also receive nilotinib hydrochloride monohydrate PO on days 7, 8, 14, and 15 of cycle 1 and days -1, 1, 7, 8, 14, and 15 of cycle 2. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Nilotinib: Given PO
  Nilotinib Hydrochloride Monohydrate: Given PO on cycle 1 Days 7, 14, 15 once a day 24 hours prior to the paclitaxel infusion and again 30 minutes prior to the paclitaxel infusion on days 8, 15.
  Paclitaxel: Given IV weekly on days 1, 8, 15, of every 21 days, at a starting dose of 80mg/m2
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Dose Level 1 (100mg Nilotinib) | Dose Level 2 (200mg Nilotinib) | Dose Level 3 (300mg Nilotinib)
Started | 5 | 3 | 2
Completed | 2 | 2 | 2
Not Completed | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (100mg Nilotinib) | Dose Level 2 (200mg Nilotinib) | Dose Level 3 (300mg Nilotinib) | Total
Number analyzed (Participants) | 5 | 3 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 2 | 10
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 10
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 2 | 9
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 4 | 2 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (Phase Ib)
Description: Will be classified and attributed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v)5.0 and will be summarized within and across dose levels using descriptive statistics. The overall number and percentage of patients experiencing adverse events (AEs) and toxicities will be summarized and reported as across all event types, non-hematologic AEs, hematologic AEs, and for each type. Specific focus will be in summarizing any neuropathy-related AEs by dose level and how this corresponds to our measures of OATP1B1 inhibition. All patients who have received at least one dose of the therapeutic agents will be evaluable for toxicity and tolerability.
Time Frame: Up to 6 weeks
Measure: Number; unit: Number of Events
Arm/Group | Dose Level 1 (100mg Nilotinib) | Dose Level 2 (200mg Nilotinib) | Dose Level 3 (300mg Nilotinib)
Number analyzed (Participants) | 5 | 3 | 2
Number of Events
  Anemia | 10 | 2 | 2
  Cardiac disorders - Other, specify | 1 | 0 | 0
  Ear and labyrinth disorders - Other, specify | 1 | 0 | 0
  Blurred vision | 1 | 0 | 1
  Eye pain | 1 | 0 | 0
  Watering eyes | 1 | 0 | 0
  Constipation | 1 | 1 | 1
  Diarrhea | 4 | 0 | 4
  Gastroesophageal reflux disease | 2 | 1 | 1
  Gastrointestinal disorders - Other, specify | 1 | 0 | 0
  Mucositis oral | 4 | 1 | 1
  Nausea | 3 | 2 | 1
  Edema limbs | 1 | 0 | 0
  Fatigue | 4 | 2 | 3
  Localized edema | 3 | 0 | 0
  Pain | 1 | 2 | 4
  Mucosal infection | 2 | 0 | 0
  Otitis externa | 1 | 0 | 0
  Injury, poisoning and procedural complications - Other, specify | 1 | 0 | 0
  Alkaline phosphatase increased | 1 | 0 | 0
  Lymphocyte count decreased | 2 | 1 | 3
  Neutrophil count decreased | 5 | 0 | 0
  White blood cell decreased | 4 | 0 | 2
  Anorexia | 4 | 0 | 0
  Hyperglycemia | 3 | 3 | 2
  Hyperphosphatemia | 1 | 0 | 0
  Arthralgia | 1 | 1 | 0
  Bone pain | 1 | 1 | 0
  Musculoskeletal and connective tissue disorder - Other, specify | 1 | 0 | 0
  Myalgia | 3 | 0 | 0
  Dysgeusia | 2 | 0 | 0
  Headache | 4 | 1 | 1
  Nervous system disorders - Other, specify | 1 | 0 | 0
  Paresthesia | 1 | 1 | 4
  Peripheral sensory neuropathy | 5 | 1 | 0
  Anxiety | 1 | 1 | 1
  Depression | 3 | 1 | 1
  Insomnia | 1 | 1 | 0
  Allergic rhinitis | 4 | 0 | 0
  Dyspnea | 2 | 1 | 3
  Alopecia | 1 | 0 | 0
  Bullous dermatitis | 1 | 0 | 0
  Nail changes | 1 | 0 | 0
  Pain of skin | 1 | 0 | 0
  Palmar-plantar erythrodysesthesia syndrome | 2 | 1 | 0
  Rash maculo-papular | 1 | 0 | 3
  Skin and subcutaneous tissue disorders - Other, specify | 5 | 0 | 0
  Flushing | 1 | 0 | 0
  Hot flashes | 1 | 0 | 0
  Hypertension | 1 | 1 | 0
  Dry mouth | 0 | 1 | 0
  Alanine aminotransferase increased | 0 | 1 | 1
  Aspartate aminotransferase increased Aspartate aminotransferase increased | 0 | 1 | 0
  Weight loss | 0 | 1 | 0
  Hypokalemia | 0 | 1 | 0
  Dizziness | 0 | 1 | 0
  Neuralgia | 0 | 1 | 0
  Peripheral motor neuropathy | 0 | 1 | 0
  Dry skin | 0 | 1 | 1
  Dysuria | 0 | 1 | 0
  Pruritus | 0 | 1 | 0
  Skin hyperpigmentation | 0 | 1 | 0
  Tinnitus | 0 | 0 | 1
  Abdominal pain | 0 | 0 | 1
  Vomiting | 0 | 0 | 4
  Breast infection | 0 | 0 | 2
  Platelet count decreased | 0 | 0 | 2
  Back pain | 0 | 0 | 1
  Joint range of motion decreased | 0 | 0 | 1
  Muscle cramp | 0 | 0 | 1
  Scoliosis | 0 | 0 | 1
  Extrapyramidal disorder | 0 | 0 | 1
  Sleep apnea | 0 | 0 | 1

2. Primary Outcome: Recommended Phase II Dose (RP2D) of Nilotinib in Combination With Paclitaxel (Phase Ib)
Description: The RP2D will be derived from an adaptive Bayesian method for dose-finding based on trade-offs between the probabilities of treatment efficacy and toxicity. In this design, treatment efficacy is defined as significant inhibition of OATP1B1 activity by nilotinib, without causing changes in the pharmacokinetic profiles of paclitaxel. Efficacy in this setting will be OATP1B1 inhibition as defined by a >= 5-fold increase in the area under the curve (AUC) of GCDCA-S from pre- to post-treatment and/or detectable CDCA-24G levels post-treatment.
Time Frame: Up to 6 weeks
Population: The 6 participants who completed study treatment were evaluated for this outcome.
Measure: Number; unit: milligrams
Groups:
- Treatment (All Phase 1b Dose Levels): Patients receive paclitaxel IV on days 1, 8, and 15. Patients also receive nilotinib hydrochloride monohydrate PO on days 7, 8, 14, and 15 of cycle 1 and days -1, 1, 7, 8, 14, and 15 of cycle 2. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Nilotinib: Given PO
  Nilotinib Hydrochloride Monohydrate: Given PO on cycle 1 Days 7, 14, 15 once a day 24 hours prior to the paclitaxel infusion and again 30 minutes prior to the paclitaxel infusion on days 8, 15.
  Paclitaxel: Given IV weekly on days 1, 8, 15, of every 21 days, at a starting dose of 80mg/m2
  Questionnaire Administration: Ancillary studies
Arm/Group | Treatment (All Phase 1b Dose Levels)
Number analyzed (Participants) | 6
milligrams | NA — A recommended phase 2 dose was not determined as none of the dose level cohorts reached the efficacy threshold.

3. Other Pre Specified Outcome: Evaluate Effects of Nilotinib and Paclitaxel (Phase Ib) on Patients Through Pharmacokinetics (PK) for Clinical Significant Interactions.
Description: Will explore PK endpoints Area under the plasma concentration versus time curve (AUC)
Time Frame: : Pre-dose, prior to starting paclitaxel (day 1, day 8), prior to starting nilotinib (day 8 only), immediately prior to end of paclitaxel, after paclitaxel on days 1 and 8 and pre-dose, after nilotinib on day 7.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/3 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=5) | Dose Level 2 (N=3) | Dose Level 3 (N=2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=5) | Dose Level 2 (N=3) | Dose Level 3 (N=2)
Anemia (Blood and lymphatic system disorders) | 2 (10) | 1 (2) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 2 (2) | 2 (3)
Localized edema (General disorders) | 2 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 2 (4)
Mucosal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (1) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (5) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (4) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 2 (3) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04205903/Prot_SAP_000.pdf
  • Informed Consent Form: Dose Dense Paclitaxel (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04205903/ICF_001.pdf
  • Informed Consent Form: Weekly Paclitaxel (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04205903/ICF_002.pdf